CLINICAL TRIAL: NCT06153433
Title: Clinical Trial to Evaluate the Efficacy and Safety of Suvaro®OD Tablet in Patients With Dyslipidemia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 4-2023-0589
Record Dates: First submitted 2023-11-22; First posted 2023-12-01 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Dyslipidemia
Keywords: dyslipidemia; orally disintegrating tablet; odt; rosuvastatin; preference
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rosuvastatin IR Tablet (Active Comparator): Rosuvastatin Immediate-Release Tablet (IRT) 10mg
  Interventions: Drug: Rosuvastatin Immediate-Release Tablet (IRT) 10mg
- SUVARO®OD Tablet (Experimental): Rosuvastatin orally disintegrating tablet (SUVARO®ODT) 10mg
  Interventions: Drug: Rosuvastatin orally disintegrating tablet (SUVARO®ODT) 10mg

INTERVENTIONS:
Drug: Rosuvastatin Immediate-Release Tablet (IRT) 10mg — Rosuvastatin Immediate-Release Tablet (IRT) 10mg
  Arms: Rosuvastatin IR Tablet
Drug: Rosuvastatin orally disintegrating tablet (SUVARO®ODT) 10mg — Rosuvastatin orally disintegrating tablet (SUVARO®ODT) 10mg
  Arms: SUVARO®OD Tablet

SUMMARY:
The aim of study is to evaluate the efficacy and safety of the new generic formulation (rosuvastatin orally disintegrating tablet (SUVARO®ODT) in patients with dyslipidemia.

DETAILED DESCRIPTION:
STUDY OBJECTIVES: The aim of study is to evaluate the efficacy and safety of the new generic formulation (rosuvastatin orally disintegrating tablet (SUVARO®ODT) in patients with dyslipidemia. Also, this study is designed to observe patients' preference and adherence for SUVARO®ODT.

HYPOTHESIS: We hypothesized that there will be no difference in LDL-C lowering efficacy of the two formulations (SUVARO®ODT 10-mg or rosuvastatin Immediate-release tablet (IR) 10-mg).

STUDY DESIGN: This is a randomized, multicenter, open-label, two-period crossover study with 112 enrolled patients.

Subjects: Patients with dyslipidemia over 50 years of age who received statin treatmen for at least 2 months

ELIGIBILITY:
Inclusion Criteria:

1. Patients with dyslipidemia over 50 years of age who received statin treatmen for at least 2 months
2. Written informed consent to participate in the trial

Exclusion Criteria:

1. History of previous hypersensitivity reaction to other statins, including rosuvastatin
2. patients with acute arterial disease within 3 months
3. Uncontrolled Hypertensive Patients defined as SBP ≥180 mm Hg and DBP ≥110 mm Hg, respectively
4. Uncontrolled diabetes mellitus (HbA1c > 9%)
5. Uncontrolled hypothyroidism defined as TSH >1.5 within the last 6 months
6. Taking other lipid lowering agent except statins
7. History of statin-induced myopathy, rhabdomyolysis
8. Patients with severe hepatic or renal dysfunction
9. BMI (body mass index) > 40 kg/m2
10. history of galactose intolerance, Lapp lactose deficiency, or glucose-galactose malabsorption

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2023-11-06 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Change in LDL-C level from Baseline after treatment of each formulation for 8 week | Week 0, 8, 16

SECONDARY OUTCOMES:
Change in Total Cholesterol (TC) from Baseline after treatment of each formulation for 8 week | Week 0, 8, 16
Change in High-density lipoprotein (HDL) from Baseline after treatment of each formulation for 8 week | Week 0, 8, 16
Change in Triglycerides (TG) from Baseline after treatment of each formulation for 8 week | Week 0, 8, 16

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Sun Kim, Principal Investigator — Division of Cardiology, Department of Internal Medicine, Yonsei Univerisity
Locations (1):
- Division of Cardiology, Department of Internal Medicine, Yonsei Univerisity,, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Olsson AG, Pears J, McKellar J, Mizan J, Raza A. Effect of rosuvastatin on low-density lipoprotein cholesterol in patients with hypercholesterolemia. Am J Cardiol. 2001 Sep 1;88(5):504-8. doi: 10.1016/s0002-9149(01)01727-1. PMID 11524058
- [Background] Zhang L, Zhang S, Yu Y, Jiang H, Ge J. Efficacy and safety of rosuvastatin vs. atorvastatin in lowering LDL cholesterol : A meta-analysis of trials with East Asian populations. Herz. 2020 Sep;45(6):594-602. doi: 10.1007/s00059-018-4767-2. Epub 2018 Nov 27. PMID 30483816
- [Background] Park JS, Kim YJ, Choi JY, Kim YN, Hong TJ, Kim DS, Kim KY, Jeong MH, Chae JK, Oh SK, Seong IW. Comparative study of low doses of rosuvastatin and atorvastatin on lipid and glycemic control in patients with metabolic syndrome and hypercholesterolemia. Korean J Intern Med. 2010 Mar;25(1):27-35. doi: 10.3904/kjim.2010.25.1.27. Epub 2010 Feb 26. PMID 20195400